CLINICAL TRIAL: NCT02549183
Title: Evaluation of Stimulation Pulse Rate on Clinical Outcomes in Patients Whose Pain is Controlled by 10KHz Frequency - a Feasibility Study
Brief Title: Evaluation of Spinal Cord Stimulation Pulse Rate On Clinical Outcomes
Acronym: PROCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: North Bristol NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B726
Record Dates: First submitted 2015-09-01; First posted 2015-09-15 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Back Pain; Neuralgia
Keywords: Spinal Cord Stimulation
MeSH Terms: conditions — Back Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator): Boston Scientific PRECISION Spinal Cord Stimulator System with MultiWave Technology programmed to A KHz
  Interventions: Device: Boston Scientific PRECISION Spinal Cord Stimulator System
- Arm 2 (Active Comparator): Boston Scientific PRECISION Spinal Cord Stimulator System with MultiWave Technology programmed to B KHz
  Interventions: Device: Boston Scientific PRECISION Spinal Cord Stimulator System
- Arm 3 (Active Comparator): Boston Scientific PRECISION Spinal Cord Stimulator System with MultiWave Technology programmed to C KHz
  Interventions: Device: Boston Scientific PRECISION Spinal Cord Stimulator System
- Arm 4 (Active Comparator): Boston Scientific PRECISION Spinal Cord Stimulator System with MultiWave Technology programmed to D KHz
  Interventions: Device: Boston Scientific PRECISION Spinal Cord Stimulator System

INTERVENTIONS:
Device: Boston Scientific PRECISION Spinal Cord Stimulator System — Spinal cord stimulation randomly programmed to KHz frequencies; A, B, C and D Kilo Hertz.

SUMMARY:
Clinical study to estimate the optimal frequency for stimulation of the spinal cord to achieve relief from back pain.

DETAILED DESCRIPTION:
This is a feasibility study to identify the optimal frequency for stimulation of the spinal cord to achieve maximum reduction in neuropathic back pain as measured by average Numerical rating Scale.

Twenty patients who suffer from back more than leg pain will be recruited into the study once they have satisfactory pain relief from both low and high frequency stimulations. Each patient will then receive stimulation at four different frequencies for 2-3 weeks in a random and blinded order. Their pain scores and function will be assessed using a variety of different tools. The data will then be used to estimate the optimal frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Complaint of persistent or recurrent low back pain, with or without equal or lesser leg pain, for at least 90 days prior to Screen.
2. Received at least 90 days of documented pain management care to address the primary pain complaint, prior to Screening (e.g. medication, physical therapy.)
3. No back surgery within 6 months prior to Screening.
4. Average low back pain intensity, during the position/activity, which routinely causes worst pain, of 5 or greater on a 0-10 numerical rating scale during Baseline period based on eDiary.
5. If taking prescription opioids for primary chronic pain complaint (low back and/or leg pain), must have been on a stable prescription (same drug(s) and dose(s)) 30 days prior to Screening to a total of less than 180 mg Oral Morphine equivalent
6. Willing and able to comply with all protocol-required procedures and assessments/evaluations (e.g. willing to comply with opioid prescription lock from the Baseline visit through End of Rate Randomization and protocol required stimulation parameter locks, complete daily eDiary).
7. 18 years of age or older when written informed consent is obtained.
8. If female of childbearing potential: not pregnant, as evidenced by a negative pregnancy test at Screening.
9. Subject signed a valid, IRB-approved informed consent form (ICF) provided in English.
10. Baseline Oswestry Disability Index score ≥ 20 and ≤ 80.
11. Received at least 30 per cent reduction in NRS of average low back pain intensity from Baseline during the end of Post Implant HF10 Sweet-Spot Search as recorded in the eDiary.

Exclusion Criteria:

1. Average worst leg pain intensity is greater than average worst low back pain intensity as reported during Baseline period based on eDiary.
2. Radiographic evidence of spinal instability requiring fusion.
3. Primary pain complaint of vascular origin (e.g. peripheral vascular disease).
4. Spinal pain secondary to neoplasm, infection, autoimmune disorder with spinal involvement, or a spinal metabolic disorder.
5. Any pain-related diagnosis or medical/psychological condition that, in the clinician's best judgment might confound reporting of study outcomes (e.g. pelvic pain, angina pain, chronic migraine.
6. Participating (or intends to participate) in another clinical study.
7. Terminal illness with anticipated survival 1 year.
8. Current condition associated with risk of immunocompromised that might increase risk of infection during study duration.
9. Currently on any anticoagulant medications that cannot be discontinued during perioperative period.
10. Are pregnant/lactating or not using adequate birth control.
11. Have untreated major psychiatric comorbidity, serious drug related behaviour issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Back pain relief | Three months
  Mean reported pain on Numerical Rating Scale (NRS)

SECONDARY OUTCOMES:
Leg pain relief | 3-6 months
  Mean reported pain on Numerical Rating Scale (NRS)
Patient global impression of change at end of Long-Term Follow-up | 6-9 months
  Questionnaire
Change in quality of life (EQ-5D) from Baseline Visit to end of Long-Term Follow-up | 6-9 months
  Questionnaire
Change in activities of Daily Living related to back pain disability from Baseline visit to end of Long-Term Follow-up | 6-9 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Simon Thomson, MD, Study Chair — National Health Service, United Kingdom
Locations (3):
- United Kingdom (3):
  - North Bristol NHS Trust, Bristol, Avon
  - Orsett Hospital, Orsett, Essex
  - South Tees NHS Foundation Trust, Middlesbrough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomson SJ, Tavakkolizadeh M, Love-Jones S, Patel NK, Gu JW, Bains A, Doan Q, Moffitt M. Effects of Rate on Analgesia in Kilohertz Frequency Spinal Cord Stimulation: Results of the PROCO Randomized Controlled Trial. Neuromodulation. 2018 Jan;21(1):67-76. doi: 10.1111/ner.12746. Epub 2017 Dec 8. PMID 29220121